CLINICAL TRIAL: NCT05552313
Title: Effects of Kinesio Taping With Thoracic Manipulation in Mechanical Neck Pain Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/12
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Athletic Tape; Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial which will consist of 2 groups. Experimental group will be given kinesio taping along with thoracic manipulation and conventional treatment whereas control group will be given sham kinesio taping along with thoracic manipulation and conventional treatment. Both groups will be recruited concurrently.
Who Masked: Participant
Masking Description: Control group will be given sham kinesio taping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesio taping with thoracic manipulation and conventional treatment (Experimental): experimental group will be given kinesio taping with thoracic manipulation and conventional treatment
  Interventions: Procedure: kinesio tape; Procedure: standard therapy
- sham kinesio taping with thoracic manipulation and conventional treatment (Sham Comparator): control group will be given sham kinesio taping with thoracic manipulation and conventional treatment
  Interventions: Procedure: kinesio tape; Procedure: standard therapy

INTERVENTIONS:
Procedure: kinesio tape — kinesio tape will be applied while patient is in sitting position. Y strip will be applied along C1 till T1.while patient's cervical spine is in contalateral side bending and rotation. same will be performed on the other side. on top of it, an I strip will be applied horizontly along C1 to C4. Both strips will be applied with 15% to 20% stretch.
Procedure: standard therapy — Thoracic manipulation along with conventional including Tens, stretching and strengthening exercises of entire neck musculature

SUMMARY:
Neck pain is considered one of the very common cause of musculoskeletal pain. It is 4th leading cause of disability with a prevalence ranges between 30% and 50% among general population. cervical pain is among 5 most contributing factors in causing years lived with disability. Mechanical neck pain is identified by neck pain that gets evoked by sustained neck postures, neck mobility and by the palpation of cervical muscles. diagnosis is made through history and physical examination and can be helpful in differentiating from other causes of neck pain. functional impairments suffered by mechanical neck pain patients include weakness of deep cervical flexors, because of activation of superficial cervical muscles, reduced mobility of cervical spine, development of forward head posture, altered proprioception and disturbed balance leading to functional disability and decline in health related quality of life. there are different treatment approaches that include pharmacotherapy, manual therapy, active exercises, stretching, traction and electrotherapy. physiotherapy is often the first line treatment approach for individuals with mechanical, idiopathic and insidious neck pain but manual therapy is preferred through its biomechanical and neurophysiological responses that eventually leads to reduction in pain and improved function in clinical practice.thoracic manipulation and kinesio taping has proved to be very effective in treating mechanical neck pain patients according to several studies despite of their certain limitations. this study aims at evaluating effects of kinesio taping combined with thoracic manipulation in mechanical neck pain patients.

DETAILED DESCRIPTION:
As young population and office workers are inclined towards computer work, so they tend to develop forward head posture or other muscular imbalance leading towards mechanical neck pain, so this population is considered in this study. substantial amount of evidence is available on the persisting treatment options and also on thoracic manipulation and kinesio taping, but none of them evaluated combined effects of both interventions. so this study aims at evaluating combined effects of kinesio taping and thoracic manipulation on pain, functional disability and cervical ROM in mechanical neck pain patients. if there are improved results by combining these interventions then clinicians can use them in combination for better results on their patients. moreover patients can also benefit from this study as they can get back to work early and lead towards better quality of life.

This randomized controlled trial will be conducted in Rehab OPD of fauji foundation hospital and foundation university institute of rehabilitation sciences using non probability purposive sampling. Sample size has been calculated as 30 using open epi sample size calculator. Patients with primary complaint of mechanical neck pain referred to rehab opd of FFH and patients of mechanical neck pain from fuirs will be recruited according to eligibility criteria. Participants will be briefed regarding the study objectives, study procedures, risks and benefits of treatment, voluntary participation and a right to withdraw. After taking informed consent, demographic data and baseline measurements, participants will be randomly allocateditno one of two groups using coin toss method.Control group will recieve sham kinesio taping along with thoracic manipulatio and conventional physiotherapy treatment whereas experimental group will reieve cervical kinesio taping along with thoracic manipulation and conventional physiotherapy treatment.

Group 1 (experimental group): Upper thoracic manipulation using screw thrust technique. conventional treatment would include moist heat pad for 10 minutes,Tens for 10 minutes, stretching and strenghtning of sternocliedomastoid, scalnes, deep neck flexors, suboccipitals and upper and middle fibres of trapezius. kinesio taping: kinesio tape in a Y shape is applied from C1 to T1 with 15% to 20% stretch. Another I strip is applied horizontly from C1 to C4 with 15% to 20% stretch.

Group 2 (control group): upper thoracic manipulation using screw thrust technique. conventional treatment would include moist heat pad for 10 minutes, Tens for 10 minutes, stretching and strenghtning of sternocliedomastoid, scalenes, deep neck flexors, suboccipitals and upper and middle fibres of trapezius. kinesio taping: sham kinesio tape is applied.

ELIGIBILITY:
Inclusion criteria:

* individuals aged 18-35 years, unilateral or bilateral pain in posterior neck, shoulder or cervical region when moving or on palpations.
* individuals with thoracic hypomobility.
* symptoms of duration more than 3 months.
* NPRS scoring of equal to or greater than 4 points.
* neck disability index score of 20% or above.

Exclusion criteria:

* history of neurologic signs or symptoms suggestive of nerve root involvement.
* prior cervical or thoracic spine fractures, dislocation or surgeries, spinal osteoporosis or infection, or whiplash.
* pregnancy
* any contraindication to manipulation or any tape allergy.
* hypertension

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
change in pain | 4 weeks
  pain will be measured using numeric pain rating scale. nprs is a 10 item scale. higher result shows more pain and low results show less pain.
Change in Cervical ROM: | 4 weeks.
  Cervical ROM will be measured using cervical ROM device. Cervical flexion, cervical extension, cervical right and left side bending, cervical right and left rotation. During evaluation, patient would be asked to perform all movements. Three repetitions will be recorded and the final mean error calculated between angles.
Change in Functional disability: | 4 weeks
  Functional disability will be measured using neck disability index questionnaire and it is used to assess self-rated disability in neck pain patients. It has 10 items and response to every item is rated on a 6 point scale from 0, indicating no disability and 5, indicating complete disability. The responses for every item are added for a total score that ranges between 0 and 50. Higher scores represent increased level of disability

SECONDARY OUTCOMES:
Change in Deep neck flexor endurance: | 4 weeks
  It will be measured using deep neck flexor endurance test. Patient would be supine or hook lying and will be asked to perform chin tuck in and hold his head 1 inch off the table. The mean deep neck flexor endurance hold time will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan